CLINICAL TRIAL: NCT03484871
Title: Resting-state Functional Connectivity Changes During Migraine Treatment: a Structural and Functional MRI Follow-up Study
Brief Title: Resting-state Functional Connectivity Changes During Migraine Treatment
Status: Withdrawn | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chin-Sang Chung, MD, PhD, Professor of neurology, Samsung Medical Center
Other Study IDs: 2016-04-028
Record Dates: First submitted 2016-09-27; First posted 2018-04-02 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether reduced frequency of migraine attacks are associated with signal alternation and connectivity of cerebral cortex.

DETAILED DESCRIPTION:
Patients with migraine show reduced cortical thickness in regions subserving pain processing, and it is related to increasing headache frequency. In the past, only one study has shown a reversibility consequence of chronic nociceptive transmission, which normalizes when the pain is adequately treated. However, little is known whether these changes predispose to migraine or represent the effect of repeated migraine attacks. Our region of interest is reduced frequency of migraine attacks are associated with reversibility of signal alternation and functional connectivity of cerebral cortex.

In 30 migraineurs with 8-14days with headache per months who already performed brain magnetic resonance imaging will be recruited. Treatment medications such as frovatriptan and topiramate will be used for 6 months. After 6 months, follow-up brain magnetic resonance imaging will be performed.

The primary outcome is the longitudinal changes in functional connectivity in pain-processing/modulating brain regions. The secondary outcome is following: 1)longitudinal changes in structural and morphological alterations in brain regions of pain processing; 2)structural, morphological, and functional correlates of treatment response; 3)changes in monthly migraine days, migraine frequecies, headache days, and headache frequencies after treatment; 4)responses to acute migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Women
* Aged 18-50
* Drug-naïve high frequency episodic migraineurs (8-14 attacks/m)
* Performed a baseline interictal brain MRI

Exclusion Criteria:

* Medication overuse
* Chronic pain other than migraine
* On treatment of major depression, bipolar, schizophrenia, or BDI>25

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with migraine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
functional MRI imaging changes | 6 month
  temporal changes in BOLD correlations in the regions of most significant correlation with periaqueductal grey; temporal changes in BOLD correlations in the regions of most significant correlation with anterior cingulate cortex; temporal changes in default mode network

SECONDARY OUTCOMES:
structural MRI imaging changes | 6 months
  changes in cortical thickness of anterior cingulate, amygdala, periquiductal grey, and sensorimotor cortex
Functional and structural correlates of treatment response | 6 months
  >50% reduction of monthly headache days
correlation of functional MRI changes with changes in clinical parameters | 6 months
  changes in monthly headache days
responses to acute migraine treatment | 6 months after the first visit
  the Migraine Assessment of Current Therapy (Migraine-ACT) = 4

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Sang Chung, MD, PhD, Principal Investigator — Department of Neurology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No